CLINICAL TRIAL: NCT05960838
Title: Evaluation of Functionality, Operability and Wearing Comfort of Two Multifunctional Shoulder Braces in Patients Who Underwent Shoulder Surgery
Brief Title: Ultrasling Quadrant Versus Bledsoe ARC Shoulder Brace
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The shoulder brace is being revised by the Producer
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ID OE-0108
Record Dates: First submitted 2020-10-20; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2022-11

CONDITIONS: Shoulder Injuries and Disorders
MeSH Terms: conditions — Shoulder Injuries; Disease

STUDY DESIGN:
Intervention Model Description: Each brace will be worn for either the first or second half (2 weeks) of the investigated immobilizing time of 4 week as determined by randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Invervention 1 (Experimental): Immobilization with the Ultrasling® Quadrant shoulder brace after surgical treatment.
  Interventions: Device: Ultrasling® Quadrant
- Intervention 2 (Control) (Active Comparator): Immobilization with the Bledsoe ARC® brace after surgical treatment.
  Interventions: Device: Bledsoe ARC®

INTERVENTIONS:
Device: Ultrasling® Quadrant — Immobilization with the Ultrasling® Quadrant (DJO Global Switzerland Sàrl, Ecublens, Switzerland) shoulder brace after surgical treatment
  Arms: Invervention 1
Device: Bledsoe ARC® — Immobilization with the Bledsoe ARC® (Breg Inc., Carlsbad, CA USA) brace after surgical treatment
  Arms: Intervention 2 (Control)

SUMMARY:
Shoulder orthoses are an essential component of both, postoperative care as well as a range of conservative treatment concepts, and thus influence the functional outcome of a wide spectrum of glenohumeral pathologies. Therefore it is important to look at them in greater detail.

A new concept, designed by DJO Global in the "Ultrasling Quadrant®" orthosis now immobilizes only the glenohumeral joint, while giving the possibility of elbow movement. It also allows multiple settings concerning the position of the glenohumeral joint like internal rotation as well as neutral or external rotation. It is yet to be seen how these changes will influence the outcome of therapy as well as how they will change the patient's perception of the orthosis and its wearing comfort. Therefore it is planned to be compared to another multifunctional shoulder brace already established on the domestic and international market, the BledsoeARC® brace.

The primary objective is to assess if one of the investigated shoulder braces Ultrasling Quadrant® or Bledsoe Arc® is perceived by patients who received shoulder surgery as superior in terms of higher wearing comfort when worn during the post-operative immobilization period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (18 years or older)
* Presence of one of the following defined shoulder pathologies with the corresponding surgical treatment:
* Patients with isolated supraspinatus repairs in double row technique with or without biceps Treatment
* Recurrent anterior instability without significant bone loss and arthroscopic Bankart repairs with three anchors
* Rockwood Type V injury treated with arthroscopic-assisted low-profile TightRope Repair plus AC-Cerclage
* Patients with rotator cuff arthropathy treated by reverse shoulder prosthesis
* Signed Informed Consent to participate in the study

Exclusion Criteria:

* Non-tolerance of one of the braces (e.g. allergy to textile component)
* Presence of concurrent pathology of the contralateral arm , that interferes with the immobilizing treatment
* Presence of another physical disability or health disorder (e.g. psychological disorders, dementia, …) that make the handling of the braces more difficult or impossible
* Patient perceived as being at risk of poor study compliance
* Occurrence of an intra-operative adverse event likely to influence the post-operative immobilization and its evaluation
* Inability to understand and speak German
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall wearing comfort subjectively reported by patients | 2 weeks
  The primary outcome for this study is the overall level of comfort as perceived subjectively by the patients themselves by a questionnaire (NRS based).

SECONDARY OUTCOMES:
Pain in ADL | 2 weeks
  Patients will report subjectively their perceived pain in achieving activities of daily living on an NRS from 0 (no pain) to 10 (maximum pain)
Difficulty | 2 weeks
  Patients will report subjectively their perceived difficulty in achieving activities of daily living on an NRS from 0 (no difficulty) to 10 (maximum difficulty)
Comfort | 2 weeks
  Patients will report subjectively their perceived comfort in achieving activities of daily living on an NRS from 0 (no comfort) to 10 (maximum comfort)
Operability | 2 weeks
  The operability is reported by the level of difficulty of handling of the braces as evaluated subjectively by the patients by a questionnaire on an NRS from 0 (no difficulty) to 10 (maximum difficulty). The patients will also be asked about the total time they wear the brace during the day.
Stability | 2 weeks
  Stability of the shoulder braces is measured with digital photographs of the braces position at different time points throughout the immobilizing time. The photographs are evaluated digitally with inserted lines that allow angle measurement. The angles of the braces position are then compared to a) the position intended to be immobilized in by the surgeon and b) the position of the brace when being worn by the patient. Differences in the in the application by the patient in comparison to the application by a professional are documented by photographs and measured digitally as well.
Compliance | 2 weeks
  Patients will be required to wear their allocated brace 24 hours a day/7 days a week, but in clinical practice the PI noted them not sticking to this routine prescription for various reasons.
  The level of compliance in wearing the braces is an essential information gained by the trial. At weekly intervals patients will be asked to report the mean time their worn the allocated or any other brace during the preceding week (0-6 hours | >6-12 hours | >12-18 hours | >18-24 hours) which allows us to draw conclusions to their compliance. The reason(s) for removing the brace will be documented.
Patient's preference for any of the two braces | 2 weeks
  At the end of the 4-week immobilization period, patients will be asked about their preference for any of the two braces including an option for undecided patients.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Schulthess Klinik, Zurich, Canton of Zurich
  - Schulthess Klinik, Zurich

IPD SHARING:
Plan to Share IPD: No